CLINICAL TRIAL: NCT04537702
Title: Prospective, Randomized Non-inferiority Trial of Streamlined Genetic Education and Testing for High-grade Epithelial Ovarian, Fallopian and Peritoneal Cancer Patients
Brief Title: Prospective Randomized Trial of Streamlined Genetic Education and Testing for Ovarian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00100538
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-07

CONDITIONS: Ovarian Cancer, Epithelial; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Intervention Model Description: Following consent, the clinical research coordinator will randomize the patient to either the Traditional Group (TG) or Streamlined Group (SG). The randomization process will have occurred previously using blocks of ten randomly computer-generated numbers. These numbers will be kept in individual, ordered envelopes. When a subject requires randomization, the next envelope in the sequence will be opened and the subject will be randomized according to the number listed in the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tradition Counseling Group (TG) (Active Comparator): After completion of baseline surveys, the TG subjects will be referred to a formal pre-test consultation with a genetic counselor. TG subjects will complete an electronic family history questionnaire (FHQ) within one week of the primary visit. A member of the genetics team will curate the results by contacting the subject to review errors and clarify any ambiguities in the pedigree. The TG subjects will then meet with the genetic counselor. After counseling, participants will be given the option to undergo a multi-gene panel genetic test. Those who agree to testing will also complete the standard genetic testing consent form. As per standard practice, patients will also be asked to provide consent for somatic tumor testing of surgical (non-cytologic) specimen. Subjects will complete a post-education distress and anxiety survey (IES) either via an email link to a confidential REDCap survey link 1-2 weeks after formal consultation.
  Interventions: Behavioral: Traditional Education
- Streamlined Group (SG) (Experimental): After completion of the baseline surveys, the SG subjects will watch an approximately eight minute long genetics education video. All subjects will then have the option to "opt out" and receive formal genetic counseling prior to making a decision about testing. If the subject elects to undergo genetic testing, she will fill out the standard genetic testing consent form. As per standard practice of the clinical genetic service at Duke Cancer Institute (DCI), patients will also be asked to provide consent for somatic tumor testing of surgical (non-cytologic) specimen. SG subjects will complete an FHQ within one week of the primary visit. A member of the genetics team will curate the results by contacting the subject to review common errors and clarify any ambiguities in the pedigree. Subjects will complete a post-education distress and anxiety survey (IES) via either an email link to a confidential REDCap survey link or over the phone 1-2 weeks after education.
  Interventions: Behavioral: Streamlined Education

INTERVENTIONS:
Behavioral: Streamlined Education — After completion of the baseline surveys, the SG subjects will watch an approximately eight minute long genetics education video. This video will be made with the assistance of Duke University genetic counselors and gynecologic oncology providers. It will consist of a discussion of genes and mutations, the recommendation of universal testing for high grade epithelial ovarian cancer, a review of genes associated with ovarian cancer predisposition, the possibility of uncertain results including variants of undetermined significance, the potential for undetected mutations in known or unknown cancer susceptibility genes, the potential impact on personal treatment and on family members, the possibility of genetic discrimination and the legal protection of genetic information.
  Arms: Streamlined Group (SG)
Behavioral: Traditional Education — The TG subjects will then meet with the genetic counselor at the previously scheduled appointment time. During this visit, they will receive approximately thirty to sixty minutes of counseling regarding genetic testing and potential results. The discussion is based on the American Society of Clinical Oncology (ASCO) and National Comprehensive Cancer Network (NCCN) guidelines of informed consent for genetic testing. After counseling, participants will be given the option to undergo a multi-gene panel genetic test either via saliva or blood sample. Those who agree to testing will also complete the standard genetic testing consent form. As per standard practice of the clinical genetic service at DCI, patients will also be asked to provide consent for somatic tumor testing of surgical specimen (non-cytologic).
  Arms: Tradition Counseling Group (TG)

SUMMARY:
Current guidelines recommend universal genetic testing for all patients with ovarian, fallopian and peritoneal cancer. The purpose of this trial is to investigate the non-inferiority of streamlined genetics education and testing for this patient population when compared to the traditional model of referral to genetic counseling. Patients will be randomized to either the streamlined or the traditional counseling arm. Those in the streamlined group will watch a brief educational video and have the option of immediate testing; The traditional counseling arm will instead be referred for a formal genetics consultation, after which they can choose to be tested. The primary outcome will be a patient reported outcome scale that assesses patient satisfaction with genetic counseling; patient anxiety and distress and cost effectiveness when using both strategies will also be evaluated. The study poses minimal risk to the patients that would not be encountered during standard of care genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* Either a) pathologically confirmed diagnosis of high-grade epithelial ovarian, fallopian or peritoneal cancer via biopsy or surgical pathology or b) cytologic diagnosis consistent with high-grade epithelial ovarian cancer.
* Presenting to Duke gynecologic oncology clinic or collaborating institution for first outpatient visit following pathologic or cytologic diagnosis. If logistic constraints prevent the patient from being enrolled at her initial visit, she will be eligible for enrollment up to initiation of her fifth cycle of chemotherapy.

Exclusion Criteria:

* Known family or personal history of an inherited cancer susceptibility mutation
* Previously received genetic counseling or testing for an inherited cancer susceptibility mutation
* Insurance provided by an insurance company that requires face-to-face genetic consultation prior to testing
* Unable to read or speak English as study design includes video assisted educational materials in English
* Blind or deaf as study design includes video assisted educational materials in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Demographic Information | Baseline
  Number of participants with children
Numeracy assessment | Baseline
  Numeracy as assessed by the Newest Vital Sign survey
Electronic Family History | Completed at least 1 week prior to genetic sample being taken
  Family cancer history up to past 3 generations
Change in anxiety and depression as measured by the IES Scale | Baseline, approximately 7 days post-education, and approximately 7 days post-results disclosure
  The Impact of Events Scale (IES) has been used widely as a means of measuring patient distress (particularly intrusive thoughts or avoidance) over a defined incident. This evaluation will be used to identify trends in anxiety or depression in both arms throughout the education and testing process. In this trial, the "incident" will be described as "the risk of my cancer being hereditary."
Distress as measured by MICRA | Approximately 7 days post-results disclosure
  The multidimensional impact of cancer risk assessment questionnaire (MICRA) is a 25-question validated tool that measures the impact of result disclosure in patients, particularly markers of distress

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Previs, MD, MS, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04537702/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04537702/ICF_001.pdf